CLINICAL TRIAL: NCT04929353
Title: (ImmunotheRapy SyMptom CApture) A RANDOMIZED CONTROLLED TRIAL OF SYSTEMATIC SYMPTOM ASSESSMENT IN CANCER PATIENTS TREATED WITH IMMUNE CHECKPOINT INHIBITORS
Brief Title: SYSTEMATIC SYMPTOM ASSESSMENT IN CANCER PATIENTS TREATED WITH IMMUNE CHECKPOINT INHIBITORS
Acronym: IRMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Of Perugia (Other)
Responsible Party: Principal Investigator, Roila Fausto, Professor of Medical Oncology at the University of Perugia, University Of Perugia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRMA
Record Dates: First submitted 2021-05-31; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Melanoma; Lung Cancer
MeSH Terms: conditions — Melanoma; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARM A (Other): Self-Reporting by electronic survey consisting of 14 items selected by the NCI-PRO-CTCAE TM ITEMS-ITALIAN (Item Library Version 1.0)
  Interventions: Other: Systematic symptom assessment
- Arm B (Other): Standard symptom reporting following the conventional modalities of clinical oncology practice
  Interventions: Other: Systematic symptom assessment

INTERVENTIONS:
Other: Systematic symptom assessment — * Systematic symptom assessment
  * Conventional symptom assessment

SUMMARY:
Immune-related adverse events (irAEs) can be different in their onset, kinetics and presentation but unlike chemotherapy are seldom predictable. Toxicity can affect nearly any organ system and multiple presentations of rare but severe irAEs have been reported, highlighting the relevance of vigilant monitoring.

Although early detection and timely management of high grade or special interest irAEs (such as cardiac and neurological) is obvious, it is unclear whether early identification of less serious events can lead to clinical benefit. Furthermore, it is of the utmost importance to develop new tools which can increase identification of side effects. The current study investigates systematic symptom assessment through an electronic patient reported outcome tool and aims to define whether this can reduce the rate of serious irAEs.

DETAILED DESCRIPTION:
Systematic collection of symptom information during immunotherapy treatment will be compared to usual care in locally advanced or metastatic lung cancer (NSCLC or SCLC) and surgically resected or advanced melanoma. Electronic survey will be administered every other day to report 14 common symptoms selected from the NCI-PRO-CTCAE TM library developed by the NATIONAL CANCER INSTITUTE (NATIONAL INSTITUTES OF HEALTH, Bethesda, Maryland) Italian version (NCI-PRO-CTCAETM ITEMS-ITALIAN-Item Library Version 1.0).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old at time of signing Informed Consent Form
* Histologically documented diagnosis of locally advanced or metastatic lung cancer (NSCLC or SCLC), surgically resected or advanced melanoma
* Patients eligible for immunotherapy in any line of treatment, either alone or in combination with other immunotherapy drugs or with chemotherapy
* Signed Informed Consent Form
* Life expectancy ≥3 months
* ECOG Performance Status of ≤2
* Adequate hematologic and end-organ function, defined by laboratory test result by investigator's judgment
* Viral hepatitis screening:

  1. Negative hepatitis B surface antigen (HBsAg) test
  2. For patients with positive total HBcAb test, hepatitis B virus (HBV) DNA test is required
  3. For patients with positive HCV antibody test, hepatitis C virus (HCV) RNA test is required

Exclusion Criteria:

* Patients receiving immunotherapy at time of enrollment
* > 1 grade adverse events from previous treatments
* Any uncontrolled symptom
* Clinically unstable brain metastases (i.e., symptomatic, not treated with RT and rapidly evolving)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2021-06-20 (Estimated); Primary Completion 2023-06-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
1. Decrease rate of irAEs ≥ grade 3 according to CTCAEs (Common Terminology Criteria for Adverse Events) with systematic symptom assessment | 36 months
  The electronic questionnaire surveys 14 symptoms selected by the NCI-PRO-CTCAE TM ITEMS-ITALIAN (Item Library Version 1.0). The patient will rate their symptoms on a 5-point ordinal scale concerning the symptom frequency (never / rarely / sometimes / often / almost always), intensity (not at all / a little / quite / a lot / very much) and sometimes their interference with usual/daily activities (not at all / a little / quite / a lot / very much). The questionnaire must be collected from all patients (ARM A and ARM B) after randomization and before first treatment administration. Patients enrolled in ARM A must answer the questionnaire every other day. Alert will then be triggered when symptom level is not within the designated range. Following every activated alert, a physical examination and biochemical blood tests must be carried out.

SECONDARY OUTCOMES:
1. Duration of irAEs ≥ grade 3 | 36 months
  Duration of irAEs ≥ grade 3
2. Emergency hospital admission | 36 months
  Emergency hospital admission
3. Admission to and duration of hospitalization | 36 months
  Admission to and duration of hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Oncologia Medica, Azienda Ospedaliera Universitaria, Perugia, PG, Italy

IPD SHARING:
Plan to Share IPD: No